CLINICAL TRIAL: NCT06417099
Title: Therapeutic Efficacy of Dihydroartemisinin in Patients With Polycystic Ovary Syndrome
Brief Title: Efficacy of Dihydroartemisinin for Treating PCOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-115(2)
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — artenimol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dihydroartemisinin Treatment Arm (Experimental): The subjects take dihydroartemisinin, 40mg tid for 90 days
  Interventions: Drug: Dihydroartemisinin

INTERVENTIONS:
Drug: Dihydroartemisinin — dihydroartemisinin 40mg tid po for 90 consecutive days

SUMMARY:
The primary research hypothesis of this study is that dihydroartemisinin is effective in restoration of regular menstrual cycles of PCOS subjects who meet at least two of three Rotterdam Criteria. Secondary research hypotheses include: dihydroartemisinin is also effective in reducing androgen, total immature follicles, and anti-Mullerian hormone.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common reproductive endocrine metabolic disorder caused by genetic and environmental factors. Artemisinin has been widely used as a first-line antimalarial drug in routine clinical practice. In recent years, artemisinin has also been reported to have significant anti-inflammatory, anti-tumor and immune-modulating effects. Our recent study revealed that artemisinin derivatives protect against PCOS development by inhibiting ovarian androgen production. Consistently in a small pilot study, dihydroartemisinin effectively reduced androgen levels, reduced immature follicles, and improved the estrous cycle in PCOS patients who strictly met all the three Rotterdam Criteria, namely hyperandrogenism, ovulation dysfunction, and polycystic ovaries on ultrasound. Nevertheless, clinical diagnosis of PCOS can be established as long as a patient fulfill two of the three Rotterdam Criteria. The present study aims to explore the therapeutic effects of dihydroartemisinin in patients with PCOS who met at least two of three (≥2) Rotterdam Criteria.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-28kg/M2
* No plan for pregnancy in the coming 6 months
* Patients should meet two of the three following criteria:

  1. Irregular cycles and ovulatory dysfunction: < 21 or > 35 days or < 8 cycles per year; > 90 days for any one cycle
  2. Polycystic ovaries: ≥12 follicles in at least one of two ovaries (diameter<10mm), confirmed by ultrasound.
  3. Elevated androgen levels: total testosterone>1.67 nmol/L.

Exclusion Criteria:

* Pregnancy.
* Patients with other endocrine diseases that can cause secondary PCOS, including but not limited to: 21 hydroxylase deficiency, prolactinoma, hypothyroidism, Cushing's syndrome, etc.
* Patients with other serious diseases affecting heart, liver, kidney, or other major organs.
* Patients with any type of cancer.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Recovery of regular menses | 180 days
  Record of vaginal bleeding within 6 months after start taking dihydroartemisinin

SECONDARY OUTCOMES:
Serum anti-Mullerian hormone (AMH) | 90 days
  Serum AMH before and after 90 days of medication
Free androgen index (FAI) | 90 days
  FAI (Total testosterone in nmol/L / SHBG in nmol/L X 100) before and after 90 days of medication
Number of immature follicles | 90 days
  Total number of immature follicles measuring 2-9 mm in diameter on ultrasound before and after 90 days of medication

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No